CLINICAL TRIAL: NCT05148091
Title: A Randomized, Double-blind, Placebo-controlled Phase Ⅰ/Ⅱ Clinical Study to Evaluate the Safety, Tolerability and Immunogenicity of SCTV01C in Healthy Population Aged ≥18 Years Previously Unvaccinated Against COVID-19
Brief Title: The Safety, Tolerability and Immunogenicity of COVID-19 Vaccine (SCTV01C) in Healthy, Unvaccinated Adults
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SCTV01C-02-1
Record Dates: First submitted 2021-11-16; First posted 2021-12-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2023-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — SCTV01C vaccine; Adjuvants, Pharmaceutic; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- 18~59 yrs. low dosage (20 μg) - SCTV01C VACCINE (Experimental): 20 participants in Phase I and 120 participants in Phase II at the age of 18~59 years old will receive two doses of low dosage (20 μg/0.5mL) SCTV01C VACCINE on Day 0 and Day 28
  Interventions: Biological: SCTV01C
- 18~59 yrs. low dosage (20 μg) - Adjuvant (SCT-VA02B ) (Placebo Comparator): 4 participants in Phase I and 20 participants in Phase II at the age of 18~59 years old will receive two doses of study adjuvant (SCT-VA02B ,0.5mL) on Day 0 and Day 28
  Interventions: Other: Adjuvant
- 18~59 yrs. low dosage (20 μg) - Saline (Placebo Comparator): 4 participants in Phase I and 20 participants in Phase II at the age of 18~59 years old will receive two doses of saline (0.5mL) on Day 0 and Day 28
  Interventions: Other: Saline
- ≥60 yrs. low dosage (20 μg) - SCTV01C VACCINE (Experimental): 20 participants in Phase I and 120 participants in Phase II at the age of ≥60 years old will receive two doses of low dosage (20 μg/0.5mL) SCTV01C VACCINE on Day 0 and Day 28
  Interventions: Biological: SCTV01C
- ≥60 yrs. low dosage (20 μg) - Adjuvant (SCT-VA02B ) (Placebo Comparator): 4 participants in Phase I and 20 participants in Phase II at the age of ≥60 years old will receive two doses of study adjuvant (SCT-VA02B, 0.5mL) on Day 0 and Day 28
  Interventions: Other: Adjuvant
- ≥60 yrs. low dosage (20 μg) - Saline (Placebo Comparator): 4 participants in Phase I and 20 participants in Phase II at the age of ≥60 years old will receive two doses of saline (0.5mL) on Day 0 and Day 28
  Interventions: Other: Saline
- 18~59 yrs. high dosage (40 μg) - SCTV01C VACCINE (Experimental): 20 participants in Phase I and 120 participants in Phase II at the age of 18~59 years old will receive two doses of high dosage (40 μg/0.5mL) SCTV01C VACCINE on Day 0 and Day 28
  Interventions: Biological: SCTV01C
- 18~59 yrs. high dosage (40 μg) - Adjuvant (SCT-VA02B ) (Placebo Comparator): 4 participants in Phase I and 20 participants in Phase II at the age of 18~59 years old will receive two doses of study adjuvant (SCT-VA02B, 0.5mL) on Day 0 and Day 28
  Interventions: Other: Adjuvant
- 18~59 yrs. high dosage (40 μg) - Saline (Placebo Comparator): 4 participants in Phase I and 20 participants in Phase II at the age of 18~59 years old will receive two doses of saline (0.5mL) on Day 0 and Day 28
  Interventions: Other: Saline
- ≥60 yrs. high dosage (40 μg) - SCTV01C VACCINE (Experimental): 20 participants in Phase I and 120 participants in Phase II at the age of ≥60 years old will receive two doses of high dosage (40 μg/0.5mL) SCTV01C VACCINE on Day 0 and Day 28
  Interventions: Biological: SCTV01C
- ≥60 yrs. high dosage (40 μg) - Adjuvant (SCT-VA02B ) (Placebo Comparator): 4 participants in Phase I and 20 participants in Phase II at the age of ≥60 years old will receive two doses of study adjuvant (SCT-VA02B, 0.5mL) on Day 0 and Day 28
  Interventions: Other: Adjuvant
- ≥60 yrs. high dosage (40 μg) - Saline (Placebo Comparator): 4 participants in Phase I and 20 participants in Phase II at the age of ≥60 years old will receive two doses of saline (0.5mL) on Day 0 and Day 28
  Interventions: Other: Saline

INTERVENTIONS:
Biological: SCTV01C — A Recombinant Trimeric S Protein Vaccine against SARS-CoV-2 Alpha and Beta Variants
  Arms: 18~59 yrs. high dosage (40 μg) - SCTV01C VACCINE; 18~59 yrs. low dosage (20 μg) - SCTV01C VACCINE; ≥60 yrs. high dosage (40 μg) - SCTV01C VACCINE; ≥60 yrs. low dosage (20 μg) - SCTV01C VACCINE
Other: Adjuvant — SCT-VA02B is the adjuvant of SCTV01C VACCINE applied as one of the control in the trial
  Other Names: SCT-VA02B
  Arms: 18~59 yrs. high dosage (40 μg) - Adjuvant (SCT-VA02B ); 18~59 yrs. low dosage (20 μg) - Adjuvant (SCT-VA02B ); ≥60 yrs. high dosage (40 μg) - Adjuvant (SCT-VA02B ); ≥60 yrs. low dosage (20 μg) - Adjuvant (SCT-VA02B )
Other: Saline — Saline is used as the other control in the trial
  Arms: 18~59 yrs. high dosage (40 μg) - Saline; 18~59 yrs. low dosage (20 μg) - Saline; ≥60 yrs. high dosage (40 μg) - Saline; ≥60 yrs. low dosage (20 μg) - Saline

SUMMARY:
SCTV01C-02-1 is a randomized, double-blind, placebo controlled Phase Ⅰ/Ⅱ clinical trial of the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) recombinant bivalent trimeric S protein vaccine manufactured by Sinocelltech, Ltd. The purpose of this study is to evaluate the safety , tolerability and immunogenicity of the experimental vaccine in healthy adults aged ≥ 18 Years previously unvaccinated.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, multi-center, placebo-controlled phase Ⅰ/Ⅱ clinical trial in adults aged ≥ 18 years previously unvaccinated. The purpose of this study is to evaluate the safety , tolerability and immunogenicity of the experimental SARS-CoV-2 protein vaccine (SCTV01C). The experimental vaccine and adjuvant (one placebo) were both manufactured by Sinocelltech, Ltd., while the saline (the other placebo) was commercially purchased. A total of 752 participants will be enrolled, with 112 at phase Ⅰ, and 640 at phase Ⅱ. There will be two dosage levels (20μg and 40μg), and two age groups (18~59 years old and ≥ 60 years old ) at both Phase Ⅰ and Phase Ⅱ. All of participants will be assigned to receive two doses of experimental vaccine(20μg or 40μg) or placebo (Adjuvant or Saline) on the schedule of Day 0 and Day 28.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years old when signing ICF;
* No other anti-SARS-COV-2 vaccines (approved for marketing or registered study) have been previously administered;
* Participants can sign written ICF and voluntarily participate in the study, and can fully understand the study procedure and the risk of participating in the study,
* Participants should have the ability to read, understand and fill the vaccination record card (VRC);
* Only for participants in Phase I : Those who are clinically judged to be healthy, the results of physical examination, vital signs and laboratory tests during the screening phase are normal;
* Only for participants in Phase II: Healthy participants or participants with stable underlying diseases;
* Fertile men and women of childbearing age voluntarily agree to take effective contraceptive measures from signing ICF to 6 months after full vaccination; the pregnancy test results of women of childbearing age are negative on screening.

Exclusion Criteria:

* Presence of fever within 72 h before vaccination (axillary temperature ≥ 37.3℃), or active tuberculosis, or in the acute phase of other diseases;
* A history of severe acute respiratory syndrome (SARS), Middle East respiratory syndrome (MERS), or other coronavirus infections or illness or relevant
* A history of allergic reactions to any vaccine or drug, such as allergy, urticaria, severe skin eczema, dyspnea, laryngeal edema, and angioneurotic edema;
* A medical or family history of seizure, epilepsy, encephalopathy and psychosis;
* Immunocompromised patients suffering or suffered from immunodeficiency diseases, important organ diseases, or immune diseases, etc.;
* Long-term use of immunosuppressive or immunomodulatory drugs for 14 or more days within 6 months prior to study enrollment, or planned use of immunosuppressive or immunomodulatory drugs within 2 years after study enrollment. The use of inhaled and topical corticosteroid is permitted;
* For Phase I participants only: Previously or currently suffering from clinically significant cardiovascular diseases (except for the hypertension that can be controlled with drugs), or clinically significant disorders related to respiratory system, liver and kidney (except for light fatty liver), gastrointestinal system (except for chronic gastritis), endocrine system, blood and lymphatic system, metabolic and skeletal systems, or malignancies (except for skin basal cell carcinoma and carcinoma in-situ of cervix), that may affect the study assessment, or cause risks during the study vaccination, or interfere with the data interpretation as determined by the investigator; For Phase II participants only: Presence of severe or uncontrollable cardiovascular diseases, or severe or uncontrollable disorders related to endocrine system, blood and lymphatic system, liver and kidney, respiratory system, metabolic and skeletal systems, or malignancies (except for skin basal cell carcinoma and carcinoma in-situ of cervix);
* Contraindications for intramuscular injection or intravenous blood sampling, including thrombocytopenia and other blood coagulation disorders;
* Participants who received any immunoglobulin or blood products in the previous 3 months, or plan to receive similar products during the study;
* Participants who received other intervention investigational drugs within 1 month before the vaccination (Except for the participants in the saline control group participating in the clinical study of COVID-19 vaccine);
* Participants vaccinated with influenza vaccine within 14 days, or with other type of vaccines within 28 days before the vaccination;
* Those who donated blood or had blood loss (≥450 mL) within 3 months before the first dose vaccination or plan to donate blood during the study period;
* Those who are pregnant or breast-feeding;
* Those who plan to donate ovum or sperms during the study period;
* Those who cannot follow the study procedures, or cannot cooperate to complete the study due to planned relocation or long-term outing;
* Those unsuitable for participating in the clinical study as determined by the investigator because of other abnormalities that are likely to confuse the study results, or non-conformance with the maximal benefits of the participants;
* For Phase I participants only: those who are tested positive for hepatitis B virus (HBV), hepatitis C virus (HCV), syphilis or HIV in terms of etiology or serology; For Phase II participants only: those who are tested positive for HIV in terms of etiology or serology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
Phase I: Incidence and severity of adverse reactions (ARs) from Day 0 to Day 7 days after each dose of vaccination. | From Day 0 to Day 7 after each dose
  Incidence and severity of adverse reactions occured from Day 0 to Day 7 after each dose of vaccination.
Phase II: Geometric mean titers (GMT) and seroconversion rate of total IgG antibody (ELISA method) against the SARS-CoV-2 Alpha, Beta and Delta variants on Day 14 after the second dose of vaccination; | Day 14 after the second dose of vaccination
  IgG GMT and seroconversion rate against the SARS-CoV-2 Alpha, Beta, Delta variants on Day 14 after the second dose of vaccination.
Phase II: GMT and seroconversion rate of neutralizing antibody (Live-virus neutralization assay) against the Alpha and Beta variants of SARS-CoV-2 on Day 14 after the second dose of vaccination; | Day 14 after the second dose of vaccination
  GMT and seroconversion rate of neutralizing antibody (Live-virus neutralization assay) against Alpha and Beta variants of SARS-CoV-2 on Day 14 after the second dose of vaccination;
Phase II: GMT and seroconversion rate of neutralizing antibody (Pseudovirus neutralization assay) against the SARS-CoV-2 Alpha and Beta variants on Day 14 after the second dose of vaccination; | Day 14 after the second dose of vaccination
  GMT and seroconversion rate of neutralizing antibody (Pseudovirus neutralization assay) against the SARS-CoV-2 Alpha and Beta variants on Day 14 after the second dose of vaccination;
Phase II: Incidence and severity of solicited AEs from Day 0 to Day 7 after each dose of vaccination; | Day 0 to Day 7 after each dose of vaccination
  Incidence and severity of solicited AEs from Day 0 to Day 7 after each dose of vaccination

SECONDARY OUTCOMES:
Phase I: GMT and seroconversion rate of total IgG antibody (ELISA method) against the Alpha, Beta, Delta variants SARS-CoV-2 and T4-Foldon on Day 28 after the first dose of vaccination; | Day 28 after the first dose of vaccination
  GMT and seroconversion rate of total IgG antibody against the Alpha, Beta, Delta variants of SARS-CoV-2 and T4-Foldon on Day 28 after the first dose of vaccination
Phase I: GMT and seroconversion rate of total IgG antibody (ELISA method) against the Alpha, Beta, Delta variants of SARS-CoV-2 and T4-Foldon on Day 14, Day 28, Day 90, Day 180 and Day 365 after the second dose of vaccination; | Day 14, Day 28, Day 90, Day 180 and Day 365 after the second dose of vaccination;
  GMT and seroconversion rate of total IgG antibody against the Alpha, Beta, Delta variants of SARS-CoV-2 and T4-Foldon on Day 14, Day 28, Day 90, Day 180 and Day 365 after the second dose of vaccination
Phase I: GMT and seroconversion rate of neutralizing antibody (Pseudovirus neutralization assay) against the Alpha and Beta variants of SARS-CoV-2 on Day 14, Day 28, Day 90, Day 180 and Day 365 after the second dose of vaccination; | Day 14, Day 28, Day 90, Day 180 and Day 365 after the second dose of vaccination
  GMT and seroconversion rate of neutralizing antibody (Pseudovirus neutralization assay) against the SARS-CoV-2 Alpha and Beta variants of SARS-CoV-2on Day 14, Day28, Day 90, Day 180 and Day 365 after the second dose of vaccination;
Phase I: GMT and seroconversion rate of neutralizing antibody (Live-virus neutralization assay) against the Alpha and Beta variants of SARS-CoV-2 on Day 14, Day 28, Day 90, Day 180 and Day 365 after the second dose of vaccination; | Day 14, Day 28, Day 90, Day 180 and Day 365 after the second dose of vaccination
  GMT and seroconversion rate of neutralizing antibody (Live-virus neutralization assay) against the Alpha and Beta variants of SARS-CoV-2 on Day 14, Day 28, Day 90, Day 180 and Day 365 after the second dose of vaccination;
Phase I: Number of IFN-γ positive (characterizing Th1) and IL-4 positive (characterizing Th2) T cell subpopulations 14 days and 90 days after the second dose of study vaccination; | Day 14 and Day 90 after the second dose of study vaccination
  Number of IFN-γ positive (characterizing Th1) and IL-4 positive (characterizing Th2) T cell subpopulations 14 days and 90 days after the second dose of study vaccination;
Phase I: Incidence and severity of solicited adverse events (AEs) from Day 0 to Day 7 days after each dose of vaccination; | Day 0 to Day 7 days after each dose of vaccination
  Incidence and severity of solicited adverse events (AEs) from Day 0 to Day 7 days after each dose of vaccination.;
Phase I: Incidence and severity of all unsolicited AEs Day 0 to Day 28 after each dose of vaccination; | Day 0 to Day 28 after each dose of vaccination
  Incidence and severity of all unsolicited AEs Day 0 to Day 28 after each dose of vaccination;
Phase I: Incidence and severity of laboratory abnormalities related AEs on Day 3 after each dose of vaccination; | Day 3 after each dose of vaccination
  Incidence and severity of laboratory abnormalities related AEs on Day 3 after each dose of vaccination;
Phase I: Incidence and severity of serious adverse events (SAEs), adverse events of special interest (AESIs) and medically attended adverse events (MAAEs) within 365 days after each dose of vaccination; | within 365 days after each dose of vaccination
  Incidence and severity of serious adverse events (SAEs), adverse events of special interest (AESIs) and medically attended adverse events (MAAEs) within 365 days after each dose of vaccination;
Phase II: Incidence and severity of all unsolicited AEs Day 0 to Day 28 after each dose of vaccination; | Day 0 to Day 28 after each dose of vaccination
  Incidence and severity of all unsolicited AEs Day 0 to Day 28 after each dose of vaccination;
Phase II: Incidence and severity of SAEs, AESIs, MAAEs within 365 days after each dose of vaccination; | within 365 days after each dose of vaccination
  Incidence and severity of SAEs, AESIs, MAAEs within 365 days after each dose of vaccination;
Phase II: GMT and seroconversion rate of total IgG antibodies (ELISA method) against the Alpha, Beta and Delta variants of SARS-CoV-2 on Day 28, Day 90, Day 180 and Day 365 after the second dose of vaccination; | Day 28, Day 90, Day 180 and Day 365 after the second dose of vaccination
  GMT and seroconversion rate of total IgG antibodies against the Alpha, Beta and Delta variants of SARS-CoV-2 on Day 28, Day 90, Day 180 and Day 365 after the second dose of vaccination;
Phase II: GMT of the neutralizing antibody titer (pseudoviral neutralization assay) against the Alpha and Beta variants of SARS-CoV-2 on Day 28, Day 90, Day 180 and Day 365 after the second dose of vaccination; | Day 28, Day 90, Day 180 and Day 365 after the second dose of vaccination
  GMT of the neutralizing antibody titer (pseudoviral neutralization assay) against the Alpha and Beta variants of SARS-CoV-2 on Day 28, Day 90, Day 180 and Day 365 after the second dose of vaccination;
Phase II: GMT and seroconversion rate of neutralizing antibody (Live-virus neutralization assay) against the SARS-CoV-2 Alpha and Beta variants on Day 28, Day 90, Day 180 and Day 365 after the second dose of vaccination; | Day 28, Day 90, Day 180 and Day 365 after the second dose of vaccination
  GMT and seroconversion rate of neutralizing antibody (Live-virus neutralization assay) against the SARS-CoV-2 Alpha and Beta variants on Day 28, Day 90, Day 180 and Day 365 after the second dose of vaccination;
Phase II: GMT of neutralizing antibody titers (pseudoviral neutralization assay) on Day 14, Day 28, Day 90, Day 180 and D365 after the second vaccination for other variants, such as Delta, Lambda and Gamma, etc. | Day 14, Day 28, Day 90, Day 180 and D365 after the second vaccination
  Phase II: GMT of neutralizing antibody titers (pseudoviral neutralization assay) on Day 14, Day 28, Day 90, Day 180 and D365 after the second vaccination for other variants, such as Delta, Lambda and Gamma, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Yimin Cui, M.D., Principal Investigator — Peking University First Hospital
Locations (5):
- China (5):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, CMU, Beijing, Beijing Municipality
  - PetroChina Central Hospital, Langfang, Hebei
  - Hunan Provincial Center for Disease Control And Prevention, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang G, Zhao K, Zhao X, Cui Y, He P, Zhang T, Wang Y, Shi R, Li Y, Wang Q, Ren Y, Chen Z, Zhao X, Xie Z, Liang Y, Tian Q, Pan J, Zhang C, Han Y, Dai Y, Ni S, Zhang Y, Yang X, Fu Y, Liu D, Li J, Zhang M, Hu Z, Xie L. Sustained immunogenicity of bivalent protein COVID-19 vaccine SCTV01C against antigen matched and mismatched variants. Expert Rev Vaccines. 2025 Dec;24(1):128-137. doi: 10.1080/14760584.2025.2456231. Epub 2025 Jan 27. PMID 39834144
- [Derived] Wang G, Zhao K, Han J, Hu Z, Zhang T, Wang Y, Shi R, Li Y, Song Q, Du H, He P, Xu S, Yang X, Fu Y, Cui Y, Xie L. Safety and immunogenicity of a bivalent SARS-CoV-2 recombinant protein vaccine, SCTV01C in unvaccinated adults: A randomized, double-blinded, placebo-controlled, phase I clinical trial. J Infect. 2023 Feb;86(2):154-225. doi: 10.1016/j.jinf.2022.11.008. Epub 2022 Nov 17. No abstract available. PMID 36403700